CLINICAL TRIAL: NCT02049879
Title: Quantification of Daily Physical Activity After an Intra-articular Corticosteroid Injection in Patients With Knee Osteoarthritis
Brief Title: Daily Activity After Corticosteroids Injection Among Knee Osteoarthritis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Philippe Corbeil, Professor, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INF-2010
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Injection (Experimental): Corticosteroids injection
  Interventions: Drug: Corticosteroids injection

INTERVENTIONS:
Drug: Corticosteroids injection — A solution of triamcinolone 40 mg (Kenalog) mixed with 3 cc of 2% xylocaine without epinephrine.

SUMMARY:
The objective of this study was to objectively measure daily physical activity and spatiotemporal gait pattern, as well as improvements in self reported symptoms and quality of life, before and six weeks after an intra-articular corticosteroids injection in patients suffering from knee osteoarthritis. Fourteen patients with unilateral knee osteoarthritis were recruited. The intra-articular corticosteroid injection was given at the end of the second week. Physical activity was objectively measured by an accelerometer worn by the participants for eight weeks. In addition, the Western Ontario and McMaster Universities Arthritis Index (WOMAC), the Medical Outcome Study Short Form-36 (MOS-SF36) and gait trials were completed every two weeks to assess symptoms, quality of life and spatiotemporal parameters of gait.

ELIGIBILITY:
Inclusion Criteria:

* 50 years old or more
* Medial knee osteoarthritis (Kellgren & Lawrence Grade I to III)

Exclusion Criteria:

* Intra-articular injection during the last six months
* Isolated femoro-patellar arthritis
* Rheumatoid arthritis
* Knee instability
* Spinal stenosis
* Lower limb fracture over the last year
* Lower limb surgery in the last three months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in Knee pain | Change from Baseline at 2, 4 and 6 weeks
Change in physical activity | Change from baseline at 2, 4 and 6 weeks

SECONDARY OUTCOMES:
Change in function and quality of life | Change from baseline at 2, 4 and 6 weeks
  Assessment with WOMAC and MOS-SF36 questionnaires
Change in Spatiotemporal gait parameters | Change from Baseline at 2, 4 and 6 weeks
  Gait symmetry was verified with regards to the swing and stance phase durations and step length

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Corbeil, PhD, Study Director — Laval University; Yoann Dessery, MSc, Principal Investigator — Laval University; Étienne Belzile, MD, Study Director — Laval University
Locations (1):
- Pavillon de l'Éducation Physique et des Sports - Université Laval, Québec, Quebec, Canada

REFERENCES:
- [Derived] Dessery Y, Belzile EL, Turmel S, Dore J, Diallo B, Corbeil P. Modulation of physical activity to optimize pain sensation following an intra-articular corticosteroid injection in patients with knee osteoarthritis. ScientificWorldJournal. 2014;2014:209165. doi: 10.1155/2014/209165. Epub 2014 Nov 16. PMID 25478585